CLINICAL TRIAL: NCT01051102
Title: A Trial Investigating the Pharmacodynamic Properties of NN5401 in Japanese Subjects With Type 1 Diabetes
Brief Title: Effect of NN5401 in Japanese Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1983; U1111-1112-3698 (Other: WHO)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Single dose of 0.5 U/kg body weight injected s.c. (under the skin)
  Arms: IDegAsp
Drug: biphasic insulin aspart 30 — Single dose of 0.5 U/kg body weight injected s.c. (under the skin)
  Arms: BIAsp 30

SUMMARY:
This trial is conducted in Japan. The aim of this clinical trial is to investigate the blood sugar lowering effect of NN5401 (insulin degludec/insulin aspart (IDegAsp)) in Japanese subjects with type 1 diabetes. Each subject will be randomised to one of the two possible treatment sequences (NN5401 followed by biphasic insulin aspart (BIAsp) 30 or biphasic insulin aspart 30 followed by NN5401).

ELIGIBILITY:
Inclusion Criteria:

* Japanese subject
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index (BMI): 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Loss of more than 400 mL blood (inclusive) in total with in the last 12 weeks or more than 200 mL blood (inclusive) in total within the last 4 weeks prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes (not inclusive 5) or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Area under the Glucose Infusion Rate curve after a single dose | From 4-12 hours

SECONDARY OUTCOMES:
Area under the insulin aspart concentration-time curve after a single dose | From 0-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Ikushima I, Hirao K, Sasaki T, Fumiaki K, Clauson P, Roepstorff C, Haahr HL. Glucose lowering effect of IDegAsp in Japanese subjects with type 1 diabetes. 56th Annual Meeting of the Japan Diabetes Society (JDS) 2013; Country: Japan City: Kumamoto
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com